CLINICAL TRIAL: NCT03791762
Title: Incidence of Postoperative Pain After Root Canal Preparation Using Three Different Instrumentation System Manufactured From Different Ni-Ti Alloys
Brief Title: Incidence of Postoperative Pain After Root Canal Preparation Using Three Different Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cangül Keskin, Doctor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK/389
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; WaveOne Gold; Reciproc Blue; ProTaper Next
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WaveOne Gold (Experimental): Root canal preparation with WaveOne Gold instrumentation system in a reciprocating manner
  Interventions: Procedure: WaveOne Gold
- Reciproc Blue (Experimental): Root canal preparation with Reciproc Blue instrumentation system in a reciprocating manner
  Interventions: Procedure: Reciproc Blue
- ProTaper Next (Experimental): Root canal preparation with ProTaper Next instrumentation system in a rotating manner
  Interventions: Procedure: ProTaper Next

INTERVENTIONS:
Procedure: WaveOne Gold — WaveOne Gold was operated by an endomotor (VDW Gold, Munich, Germany) at "WaveOne ALL" setting.
  Other Names: Reciprocating root canal preparation instruments; Dentsply Sirona, Ballaigues, Switzerland
  Arms: WaveOne Gold
Procedure: Reciproc Blue — Reciproc Blue was operated by an endomotor (VDW Gold, Munich, Germany) at "Reciproc ALL" setting.
  Other Names: Reciprocating root canal preparation instruments; VDW, Munich, Germany
  Arms: Reciproc Blue
Procedure: ProTaper Next — ProTaper Next was operated by an endomotor (VDW Gold, Munich, Germany) with 16:1 contra angle at the settings suggested by the manufacturer (350 rpm, 3 Ncm).
  Other Names: Rotating root canal preparation instrument; Dentsply Sirona, Ballaigues, Switzerland
  Arms: ProTaper Next

SUMMARY:
In an ideal endodontic treatment, maintenance of the original root canal morphology of the canal during root canal preparation, an ideal preparation and obturation is essential. Even if all stages are ideal, pain after endodontic treatment is a clinical condition that may occur after a few hours or several days. Post-operative pain after endodontic treatment is an undesirable condition which makes the clinician and the patient a distressing condition. Many clinical studies reported a 25-40% postoperative pain rate after endodontic treatment, which means that postoperative pain is a clinical symptom that should be considered for endodontist.

The ProTaper Next files (Dentsply Tulsa Dental Specialties) operate in continuous rotary motion, and their center of mass or center of rotation is positioned off-center relative to the instrument's central axis of rotation. During rotation, the files of this design produce a mechanical wave of motion, which travels along the length of the working part of the instrument, minimizing the contact between the file and dentin. According to the manufacturer, the offset design of this instrument also improves debris removal and flexibility in the working part of the file.

New heat treatment has been carried out on NiTi alloy, seeking to increase its flexibility and cyclic fatigue resistance. Recently, the Wave One Gold instrument, manufactured with a new thermal treatment called Gold treatment, was introduced on the market presenting some differences in design, size and taper compared to Wave One. Wave One Gold instrument has a parallelogram cross-sectional design, having two cutting edges, and consists of four instruments, 21/.06 (small), 25/07 (primary), 35/06 (medium) and 45/05 (large) while Wave One presents convex triangular cross-sectional design, besides larger size and taper.

Reciproc blue (REB, VDW), a new-generation reciprocating single-file system, is the latest version of REC. Like the REC file, REB also has an S-shaped cross section, 2 cutting edges, and a noncutting tip. However, REB files are manufactured by altering the molecular structure through a new heat treatment in order to increase the cyclic fatigue resistance. This new heat treatment gives the file its blue color. It was reported that REB files have approximately 2 times higher cyclic fatigue resistance than REC files. In addition, REB files can also be relatively prebent to better access curved canals.

However, the effect of Reciproc Blue, Protaper Next, Waveone Gold within preparation on the postoperative endodontic pain has not been investigated, yet. The aim of this prospective clinical trial was to clinically compare the incidence of postoperative pain after use of different nickel titanium file systems. The purpose of the present study was to evaluate the incidence of postoperative pain root canal preparation performed with Reciproc Blue, Protaper Next, Waveone Gold. The null hypothesis tested was that there is no difference in the incidence and severity of postoperative pain following with any of the 3 instruments.

DETAILED DESCRIPTION:
In the study, 180 patients who were diagnosed with asymptomatic irreversible pulpitis, symptomatic irreversible pulpitis, acute apical periodontitis and chronic apical periodontitis, and who applied to the Endodontics clinic for inclusion in the endodontics clinic will be included. A female with systemic healthy patients who meet the inclusion criteria will be treated clinically and radiologically. The age and gender of the patient will be recorded as patient-dependent variables, and location and type of the tooth to be treated will be recorded as tooth-dependent variables. Before the root canal treatment, the responsible researcher will provide training on patients with the Vizual Analog Scale (VAS) and its use. Root canal treatments will be completed by this responsible investigator. Before starting root canal treatment, local anesthesia will be applied using 2: Lidocaine anesthetic solution containing 2: 80,000 epinephrine using the appropriate technique to the tooth. After anesthesia is provided, endodontic access cavities suitable for the teeth will be opened. The pulp tissue will be extruded using a turner. Subsequently, according to the entry path file to be used, the subjects will be assigned to the group that is selected from the closed envelopes that write the names of the groups, and random manual preparation will be divided into 3 groups: the R-Pilot file will be used, the rotation preparation will be used, and the ProGlider file will be used (n = 60). Working lengths will be determined by using K type file 10 and electronic apex finders. The manual preparation group will serve as the control group. In this group, K type hand files (Dentsply Sirona) # 08, 10, 15, respectively, will be used with the "forward and retract" technique proposed by Ruddle at the working length. The file will be moved clockwise and then counterclockwise, by rotating quarterly, the resistance will be advanced and retracted to the point where resistance is felt in the canal. This preparation will be made with each file until the working length is reached. In the rotation group where ProGlider file will be used, the entry way will be prepared at 300 rpm and 5 Ncm torque values using the torque-controlled endodontic motor (X-Smart) until the working length is reached with the crown-down technique. In the reciprocating movement group where the R-Pilot file will be used, the entry path will be prepared using the "Reciproc All" mode in the VDW-Silver endodontic engine. After the entryway preparation, standard procedures will be performed for all three groups. The channels will be prepared with ProTaper Next file system. During treatment, 10 mL of 5% NaOCl irrigation for each channel will be done using a 30-G irrigation needle. After the preparation, final irrigation will be done with 17% EDTA, distilled water and 5% NaOCl, respectively. In the samples in all three groups, after the root canals are dried with sterile paper cone, they will be filled with cold Plus lateral compaction technique with AH Plus canal paste and gutta percha cone. Patients' phone numbers will be taken, a copy of the VAS form will be delivered to the patients to be filled in, and it will be explained that postoperative pain measurements will be made with 6, 12, 18, 24, 36 and 48 hours of VAS. Patients will be reached by phone 48 hours after the completion of root canal treatments and information about their pain levels will be received. VAS values will be classified as follows: 0, no pain; 1-3, mild pain; 4-6, moderate pain; 7-10, severe pain. The use of analgesics will also be evaluated and recorded within the first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no systemic disease or condition
* Patients having a maxillary or mandibular teeth diagnosed with one of the plural and periodontal diseases (asymptomatic irreversible pulpitis, symptomatic irreversible pulpitis, symptomatic apical periodontitis or asymptomatic apical periodontitis)

Exclusion Criteria:

* Patients, who were diagnosed with acute or chronic apical abscesses
* Patients showing signs of systemic infection
* Patients with allergies to local anesthetic agents,
* Patients who are taking medication (analgesic, antibiotic or anti-inflammatory drugs) during the 7 days before the procedure
* Patients presenting with multiple teeth requiring treatment or having a progressive periodontal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores using Visual Analogue Scale | 72 hours
  Visual analogue scale is a measure of pain intensity. In the present study, the visual analogue scale included a 10 cm straight horizontal line numbered at each centimetre from 0 to 10 showing two extreme symptoms of pain. "0" means no pain and "10" means the worst pain the subject has ever experienced. Each centimeter represents the pain intensity that the subject will mark orientated from 0 to 10. The intensity is increased from 0 to 10, therefore a higher score means a higher pain intensity and a worse outcome. 1-3 means "mild pain", 4-6 means "moderate pain" and 7-9 means "severe pain". There are no subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem Yilmaz, Samsun, Turkey (Türkiye)